CLINICAL TRIAL: NCT00916955
Title: Genetic Modifiers for 22q11.2 Syndrome
Acronym: VCFS
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Bernice Morrow, Ph.D., Albert Einstein College of Medicine
Other Study IDs: 3669FF
Record Dates: First submitted 2008-03-24; First posted 2009-06-10 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2010-08

CONDITIONS: 22q11.2 Deletion Syndrome
Keywords: 22q11.2 deletion syndrome; velo-cardio-facial syndrome; congenital anomalies; mental illness; congenital heart disease
MeSH Terms: conditions — DiGeorge Syndrome; Congenital Abnormalities; Mental Disorders; Heart Defects, Congenital | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Individuals with 22q11.2 deletions: Individuals confirmed with the diagnosis of velo-cardio-facial syndrome by positive FISH or CGH microarray confirming the diagnosis and deletion of 22q11.2
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observe development of syndrome over time

SUMMARY:
The purpose of the project is the determination of how the deletion of DNA from chromosome 22 at the q11.2 band causes the phenotypes observed in velo-cardio-facial syndrome (VCFS). In other words, the purpose remains genotype-to-phenotype matching. Current methods includes the use of whole genome chips and microarray analysis. Blood samples are collected for DNA from every patient who consents from the VCFS Center at Upstate Medical University. They are examined for phenotypic features consistent with our typical clinical evaluation. The information from these examinations will be entered anonymously into a database. Genomic information is then matched to clinical phenotype with appropriate statistical method applied.

ELIGIBILITY:
Inclusion Criteria:

* FISH confirmed diagnosis of 22q11.2 deletion syndrome

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with velo-cardio-facial syndrome confirmed by FISH
Sampling Method: Non-Probability Sample
Dates: Start 2008-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
gene signal strength | 4 years

SECONDARY OUTCOMES:
physical phenotype | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Shprintzen, PhD, Principal Investigator — Upstate Medical University; Bernice Morrow, PhD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- VCFS International Center, Syracuse, New York, United States

REFERENCES:
- [Result] Shprintzen RJ, Higgins AM, Antshel K, Fremont W, Roizen N, Kates W. Velo-cardio-facial syndrome. Curr Opin Pediatr. 2005 Dec;17(6):725-30. doi: 10.1097/01.mop.0000184465.73833.0b. PMID 16282778
- See also: Web site of the location for the investigation — http://www.vcfscenter.org